CLINICAL TRIAL: NCT01018277
Title: Effect of Mobilization on Acute Postoperative Pain and Nociceptive Function After Total Knee Arthroplasty: A Prospective, Consecutive, Trial
Brief Title: Effect of Mobilization on Acute Postoperative Pain and Nociceptive Function
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: H-1-2009-115; 2009-41-4004
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Pain, Postoperative; Pain Sensitivity, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Mobilization (walking) — 25 meters twice

SUMMARY:
Aim of the present study is twofold.

* First we want to evaluate the effect of mobilization on acute postoperative pain
* Second to test weather chances in pain sensitivity are occurring following surgery and mobilization after total knee arthroplasty

DETAILED DESCRIPTION:
Little is known about the effect of mobilization on acute postoperative pain and mobilization induced pain, and if altered pain sensitivity occur under these circumstances.

* First we want to evaluate the effect of mobilization on acute postoperative pain using the visual analog scale (VAS)
* Second to test weather chances in pain sensitivity are occurring following surgery and mobilization after total knee arthroplasty, using two simple tools, the Pain Matcher and a Pressure Algometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total unilateral knee arthroplasty

Exclusion Criteria:

* Cognitive dysfunction or peripheral / central neurological dysfunction inconsistent with protocol completing
* Alcohol and medical abuse (as defined by the National Health Service of Denmark
* Daily use of opioids or glucocorticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated with TKA
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pain score on the visual analog scale (difference before and after two mobilisation seances) | up to 24 hours
  pain at rest (supine) 5 min after exercise(after the 2nd walk)

SECONDARY OUTCOMES:
Pain score on the visual analog scale (difference before and after two mobilisation seances) | up to 24 hours
  pain at rest (supine) 20 min after the 2nd walk, pain during passive hip flexion and pain during passive knee flexion 5 and 20 min after the 2nd walk, as well as pain during the 2nd walk after 6 and 25 m
Pain sensitivity measured with pressure algometry and with pain matcher (difference before and after two mobilisation seances and difference before and after surgery) | up to 24 hours
  Nociceptive function before and after postoperative exercise

CONTACTS AND LOCATIONS:
Overall Officials: Troels Haxholdt Lunn, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark